CLINICAL TRIAL: NCT05110547
Title: Multicenter Study of Blood Biomarkers of Mitochondrial and Peroxisomal Metabolism to Differentiate Idiopathic Parkinson's Disease From Related Conditions
Acronym: BiomarPark
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MOREAU 2020
Record Dates: First submitted 2021-10-11; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Parkinson Disease; Parkinsonian Syndrome
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Parkinson's disease: patients meeting the current clinical criteria whose disorders have progressed for strictly more than 2 years and strictly less than 7 years.
  Interventions: Biological: blood collection
- atypical Parkinsonian syndromes: including the subgroups: multiple system atrophy, progressive supranuclear palsy, corticobasal degeneration with a duration of disease progression strictly greater than 2 years and strictly less than 7 years, and meeting the current clinical criteria for each
  Interventions: Biological: blood collection

INTERVENTIONS:
Biological: blood collection — 2 additional 5ml EDTA tubes, with assays for the following markers: 24S and 27 hydroxycholesterol (gas chromatography-mass spectrometry, GC-MS), Neurofilaments (SIMOA), oxydative phosphorylation (OXPHOS) and quantitative measurement of intracellular ATP (ELISA), Very long chain fatty acids (GC-MS), Octanoyl CoA (HPLC), Uric acid, MDA assay (TBAR assay kit), and Lipid panel.

SUMMARY:
With the aging of the population due to an increase in longevity, the number of people with Parkinson's disease is increasing (166,712 in France, as of December 31, 2015) and the number of patients with motor or cognitive-behavioral disorders is already a major public health challenge (1). In neurodegenerative diseases, the current strategy is to identify the disease early and, if possible, to consider therapeutic measures to slow down the progression of the disease.

Classically, when faced with the early stages of Parkinsonism, the investigators differentiate idiopathic Parkinson's disease (IPD) from atypical Parkinsonian syndromes (AP), which include multiple system atrophy (MSA), corticobasal degeneration (CBD), and progressive supranuclear palsy (PSP), for which the prognoses are more severe and the therapies less effective. In the early stage of the disease, when the symptoms are not do no yet differentiate the diseases, the differential diagnosis between IPD and PSP is a real challenge for clinicians (2). Cerebral MRI can help in the diagnosis but is most often only an indicator, as it may be normal in the early stages of the disease (2). The recent emergence of targeted therapies, specific to tauopathies or synucleinopathies, makes it essential to establish a diagnosis as early as possible in order to curb the evolution of the disease (3).

The investigators propose here a first study on the analysis of biomarkers of neurodegeneration from lipid metabolism allowing to discriminate IPD and AP from peripheral blood. Two recent studies have provided evidence of the discriminatory character of neurofilament blood testing in the early phases of parkinsonism (4,5). On the other hand, to our knowledge, none of them has studied markers from mitochondrial and peroxisomal metabolism, which could play a key role in the pathophysiology of these diseases (6,7,8,9,10).

Our strategy will therefore be to study idiopathic or atypical Parkinsonism subjects with a clearly established diagnosis in a cross-sectional manner, and to identify one or more blood markers of neurodegeneration predictive of IPD or AP, hypothesizing that these markers will be at significantly different levels between the two groups (descriptive analysis). The markers studied will include markers of neurodegeneration, markers of mitochondrial function, peroxisomal function and oxidative stress. The investigators will then study the correlations between these biomarkers and motor scores of disease severity.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Person who was informed of the study and who did not object to inclusion
* Age ≥ 18 years
* Patient affiliated to national health insurance
* Onset of symptoms strictly more than 2 years and less than 7 years ago
* Inclusion in the "NS-park" national database
* Patient with a recent brain MRI to exclude patients with secondary parkinsonism (vascular parkinson,hydrocephalus at normal pressure)

For patients in the "idiopathic Parkinson's disease group" :

- Idiopathic Parkinson's disease that is "possible," "probable," or "definite" according to UKPDSBB (UK Parkinson's Disease Society Brain Bank, Hughes et al. 1992) criteria.

For patients in the "atypical parkinsonian syndrome" group:

* Subjects with a "possible" or "probable" diagnosis of MSA according to the diagnostic criteria of Gilman et al, 2008
* Or Subjects with a "possible" or "probable" diagnosis of AP according to the diagnostic criteria of Hoglinger et al, 2017
* Or Subjects with a "possible" or "probable" diagnosis of CBD according to the diagnostic criteria of Armstrong et al, 2013

Exclusion Criteria:

For all patients:

* Disability making it impossible for him/her to participate in the trial due to lack of understanding of the information provided to him/her
* Patient under guardianship, curatorship or a measure of judicial protection
* Patients with any other neurological disease that could bias the results of our study: stroke, brain tumor, other neurodegenerative disease of the nervous system.
* Patients with secondary Parkinsonism (iatrogenic, toxic, inflammatory, post-traumatic)
* Patients with dyslipidemia receiving lipid-lowering treatment (statins, fibrates, inhibitors of intestinal cholesterol absorption).
* Patients with a progressive systemic disease that affects cholesterol metabolism, peroxisomal or mitochondrial function. (Examples: familial hypercholesterolemia, mitochondriopathy, peroxisome biogenesis disorders, etc.)
* Patient with a chronic disability making it impossible to collect clinical and cognitive data.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who regularly consult or are hospitalized at the Dijon University Hospital (in the Parkinson's disease unit) and at the Besancon University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Plasmatic measurement of 24S and 27 hydroxycholesterol | Baseline
  Markers of neurodegeneration
Plasmatic measurement on total leukocytes of the level of complexes 1 to 5 associated | Baseline
  Markers of mitochondrial function
Plasma assay of very long chain fatty acids | Baseline
  Markers of peroxisomal function:
Plasmatic measurement of ATP production | Baseline
  Markers of mitochondrial function
Plasma and leukocyte determination of Octanoyl Coenzyme A | Baseline
  Markers reflecting the relationship between peroxisome and mitochondria:
Dosage of uric acid | Baseline
  Markers of oxidative stress
Dosage of malondialdehyde (MDA) | Baseline
  Markers of oxidative stress
Plasmatic level of neurofilaments (SIMOA) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France